CLINICAL TRIAL: NCT01200758
Title: A Two-Stage Phase III, International, Multi-Center, Randomized, Controlled, Open-Label Study to Investigate the Pharmacokinetics, Efficacy and Safety of Rituximab SC in Combination With CHOP or CVP Versus Rituximab IV in Combination With CHOP or CVP in Patients With Previously Untreated Follicular Lymphoma Followed by Maintenance Treatment With Either Rituximab SC or Rituximab IV
Brief Title: A Study of Rituximab (MabThera) Subcutaneous (SC) Versus Rituximab (MabThera) Intravenous in Participannts With Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO22334; 2010-021377-36
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) (Active Comparator): Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) in combination with up to 8 cycles of cyclophosphamide, doxorubicin, vincristine, prednisolone (CHOP) or cyclophosphamide, vincristine, prednisolone (CVP) chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
  Interventions: Drug: Rituximab IV; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/Prednisolone
- Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP) (Experimental): First cycle of rituximab IV infusion (375 mg/m^2) + 7 cycles of rituximab SC (1400 mg; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
  Interventions: Drug: Rituximab SC; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: Rituximab SC — First cycle of rituximab IV infusion (375 mg/m^2) + 7 cycles of rituximab SC (1400 mg; rituximab induction) in administered every 3 weeks. Participants achieving at least PR entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
  Other Names: MabThera
  Arms: Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Drug: Rituximab IV — Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
  Other Names: MabThera
  Arms: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP)
Drug: Cyclophosphamide — Eight cycles of cyclophosphamide (750 mg/m^2 IV) administered every 3 weeks.
Drug: Doxorubicin — Eight cycles of doxorubicin (50 mg/m^2 IV) administered every 3 weeks.
Drug: Vincristine — Eight cycles of doxorubicin (1.4 mg/m^2 IV) administered every 3 weeks.
Drug: Prednisone/Prednisolone — Eight cycles of prednisone/prednisolone (100 mg/day or 40 mg/m^2/day IV/orally) administered Days 1 to 5 of every 21 days cycle.

SUMMARY:
This two-stage, multi-center, randomized, controlled, open-label study will investigate the pharmacokinetics, efficacy and safety of rituximab SC versus rituximab IV in participants with previously untreated follicular non-Hodgkin's lymphoma. Participants will be randomized to receive 375 milligrams per meter square (mg/m^2) rituximab as IV infusion or 1400 milligrams (mg) rituximab SC. In addition, participants will receive standard chemotherapy. Participants who achieved a complete or partial response (PR) after 8 treatment cycles, will receive maintenance treatment for a further maximum number of 12 cycles. Maintenance treatment cycles will be repeated every 8 weeks. This is a two-stage study. Stage 1 was designed to confirm the chosen rituximab SC dose resulting in comparable rituximab serum Ctrough levels compared with rituximab IV, when given as part of induction treatment every 3 weeks. Enrollment for Stage 2 started after the rituximab SC dose was established in Stage 1. Stage 2 aimed to further investigate the efficacy and safety of rituximab SC compared with rituximab IV. The anticipated time on study treatment is 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cluster of differentiation 20 (CD20)-positive, follicular Non-Hodgkin's lymphoma grade 1, 2, 3a. A tumor biopsy must have been performed within 6 months before study entry with material available for central review
* No prior treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Grade 3b follicular lymphoma
* Transformation to high-grade lymphoma secondary to follicular lymphoma
* Types of Non-Hodgkin's lymphoma other than follicular lymphoma
* Presence or history of central nervous system (CNS) disease
* Corticoid therapy during the last 4 weeks, except prednisone treatment less than (<) 20 milligrams per day (mg per day)
* Known active bacterial, viral, fungal, or mycobacterial, or any major episode of infections requiring hospitalization or treatment with IV antibiotics within 4 weeks of start of study medication, or oral antibiotics within 2 weeks prior to start of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2012-06-12 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (152):
- Australia (5):
  - Gosford Hospital; Cancer Care Services, Gosford, New South Wales
  - Wollongong Hospital; Cancer Services, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast Hospital; Haematology Department, Southport, Queensland
  - Queen Elizabeth Hospital; Haematology, Woodville South, South Australia
- Belgium (3):
  - UZ Antwerpen, Edegem
  - CHU Sart-Tilman, Liège
  - Sint Augustinus Wilrijk, Wilrijk
- Bosnia and Herzegovina (3):
  - University Clinical Center of the Republic of Srpska, Clinic for Internal Disease, Hematology Dept, Banja Luka
  - University Clinical Center Sarajevo, Clinic for Hematology, Sarajevo
  - University Clinical Centre Tuzla, Clinic for Oncology, Hematology and Radiotherapy, Tuzla
- Brazil (5):
  - Nucleo de Hematologia e Transplante de Medula Ossea de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Misericordia de Sao Paulo; Hematologia e Hemoterapia, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Bulgaria (4):
  - UMHAT Dr Georgi Stranski; Hematology, Pleven
  - Umhat S. George; Hematology, Plovdiv
  - Specialised Hospital For Treatment Of Hematological Diseases; Hematology, Sofia
  - Mhat Sveta Marina; Dept. of Haematology, Varna
- Canada (6):
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - Centre de sante et de services sociaux Rimouski Neigette, Rimouski, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
  - CHU de Quebec - Hopital de l'Enfant-Jesus; Unite de Recherche en Hematologie et Oncologie, Québec
- Colombia (4):
  - Fundacion Cardioinfantil, Bogotá
  - Centro Medico Imbanaco, Cali
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
  - Oncólogos de Occidente, Pereira
- Croatia (2):
  - UHC Rijeka, Rijeka
  - University Hospital Center Zagreb; Haematology Department, Zagreb
- Denmark (6):
  - Aarhus Universitetshospital, Hæmatologisk Afdeling R, Aarhus
  - Herlev Uni Hospital; Hæmatologisk Afdeling L 121, Herlev
  - Rigshospitalet; Hæmatologisk Klinik, København Ø
  - Odense Universitetshospital; Hæmatologisk Afdeling, Odense C
  - Sygehus Syd Roskilde; Onkologisk/haematologisk ambulatorium, Roskilde
  - Vejle Hospital; Dept of Medicine, Division of Hematology, Vejle
- Helsinki University Central Hospital; Dept of Oncology, Helsinki, Finland
- France (12):
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Hopital Henri Mondor; Hematologie Clinique, Créteil
  - Chu Site Du Bocage;Hematologie Clinique, Dijon
  - Clinique Victor Hugo; Chimiotherapie, Le Mans
  - Institut J Paolii Calmettes; Onco Hematologie 1, Marseille
  - Hopital Saint Eloi; Hematologie Oncologie Medicale, Montpellier
  - Hopital Hotel Dieu Et Hme;Hopital De Jour, Nantes
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - Hopital De Haut Leveque; Hematologie Clinique, Pessac
  - Ch Lyon Sud; Hemato Secteur Jules Courmont, Pierre-Bénite
  - Hopital De La Miletrie; Hematologie Et Oncologie Medicale, Poitiers
  - Hopital Bretonneau; Hematologie Therapie Cellulaire, Tours
- Georgia (4):
  - M.Zodelava's Hematology Center, Tbilisi
  - Mediclub, Tbilisi
  - Institute of Hematology and Transfusiology, Tbilisi
  - Chemotherapy and Immunotherapy Clinic Medulla, Tbilisi
- Germany (20):
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Gemeinschaftspraxis PD Dr. med. Marcel Reiser und Dr. med. Ildiko Kátay, Cologne
  - Klinikum Darmstadt GmbH; Med. Klinik V; Onkologie & Hämatologie, Darmstadt
  - Gemeinschaftspraxis Dr. med. J. Mohm und Dr. med. G. Prange-Krex; Fachaerzte fuer Innere Medizin, Dresden
  - PIOH PD Dr. R. Schnell - Dr. H. Schulz - Dr. M. Hellmann, Frechen
  - Universitätsklinikum Gießen und Marburg GmbH Standort Gießen Medizinische Klinik I, Giessen
  - Universitätsklinikum Greifswald Klinik für Innere Medizin C und Poliklinik, Greifswald
  - Internistisch-Onkologische Gemeinschaftspraxis; Dres. Rohrberg, Hurtz, Schma usw., Halle
  - Medizinische Hochschule; Zentrum Innere Medizin; Abt. Hämatologie u. Onkologie, Hanover
  - St. Vincentius Kliniken Ag; Medizinische Klinik Abt. 2, Karlsruhe
  - UKSH Klinik für Innere Medizin II, Hämatologie und Internistische Onkologie, Kiel
  - Onkologische Gemeinschaftspraxis, Magdeburg
  - Gemeinschaftspraxis Fr. Dr. med. Balser & Hr. Dr. med. Weidenbach, Marburg
  - Medizinisches Versorgungszentrum MOP, München
  - Praxis Dr.med. Jens Uhlig, Naunhof
  - Praxis Dr. Clemens Müller-Naendrup (Onkologische Schwerpunktpraxis im MVZ 2 GmbH), Olpe
  - Prosper-Hospital, Medizinische Klinik I, Recklinghausen
  - Praxis Dr. Fenchel, Saalfeld
  - Caritas Kilinik St. Theresia; Abt. Innere Medizin, Saarbrücken
  - Praxis für Hämatologie & Onkologie, Saarbrücken
- Greece (2):
  - Laiko General Hospital of Athens; A Propedeutical Clinic of Internal Medicine, Athens
  - Attiko Hospital; Haematology Clinic, Athens
- Italy (10):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Ematologia E Trapianto Di Midollo Osseo, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera Ospedale S.Carlo; Ematologia, Potenza, Basilicate
  - A.O. Universitaria Federico II Di Napoli; Oncologia Ed Endocrinologia Clinica, Napoli, Campania
  - AUSL - IRCCS Santa Maria Nuova; U.O. Day Hospital di Oncologia, Reggio Emilia, Emilia-Romagna
  - Ospedale S. Eugenio; Divisione Di Ematologia, Rome, Lazio
  - Uni Degli Studi Di Genova; 1A Divisione Di Ematologia, Genoa, Liguria
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili;U.O. Ematologia, Brescia, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Emato-Oncologia, Milan, Lombardy
  - Ospedale Ca Foncello; Ematologia, Treviso, Veneto
  - Ospedale Di Vicenza; Nefrologia, Ematologia, Vicenza, Veneto
- Malaysia (3):
  - University Malaya Medical Center; Hematology Unit of Department of Internal Medicine, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Sarawak General Hospital; Department of Radiotherapy, Oncology and Palliative care, Sarawak, Sarawak
  - Ampang Hospital; Department of Haematology, Ampang
- Mexico (4):
  - Centro Estatal De Cancerologia De Chihuahua; Servicio De Hematologia Banco De Sangre, Chihuahua City
  - Hospital General De Culiacan; Servicio De Hematologia, Culiacán
  - Hospital Universitario Dr. Jose E. Gonzalez; Haematology, Monterrey
  - Centro de Estudios Clinicos de Queretaro (CECLIQ), Querétaro
- New Zealand (2):
  - Canterbury Health Laboratories; Haematology, Christchurch
  - Palmerston North Hospital; Regional Cancer Treatment Service, Palmerston North
- North Macedonia (2):
  - University Clinic for Hematology; HSCT Department, Skopje
  - University Clinic of Hematology Skopje, Hospital Care Department, Skopje
- Peru (3):
  - Instituto;Oncologico Miraflores, Lima
  - Oncosalud Sac; Oncología, Lima
  - Hospital Maria Auxiliadora, Lima
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Brasov,Clinica de Hematologie, Brasov
  - Fundeni Clinical Inst. ; Hematology Dept, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Spiridon Iasi, Clinica de Hematologie, Iași
  - Institutul Regional de Oncologie Iasi; Clinica de Hematologie, Iași
  - Spitalul Clinic Judetean de Urgenta Targu-Mures; compartiment Hematologie, Târgu Mureş
  - Spitalul Clinic municipal de Urgenta Timisoara; Clinica de Hematologie, Timișoara
- Russia (7):
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - Haematology Research Center; Haematology, Moscow
  - Penza Regional Oncology Dispensary, Penza
  - Research Inst. of Hematology & Blood Transfusion ; Hematology, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov; Hematology, transfusiology and transplanta, Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies; Dept of Radiology, St.Petersburg, Pesochny
- Serbia (2):
  - Institute of Hematology, Belgrade
  - Clinical Center Vojvodine; Clinic for Hematology, Novi Sad
- Singapore (3):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - Singapore General Hospital; Department of Haematology, Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- Slovakia (2):
  - St. Elisabeths Cancer Center, Bratislava
  - National Cancer Inst. ; Dept. of Chemotherapy, Bratislava
- South Africa (5):
  - National Hospital; Oncotherapy Dept, Bloemfontein
  - Durban Oncology Center, Durban
  - University of Witwatersrand/Johannesburg Hospital; Dept. of ocnology, Johannesburg
  - Cancercare, Kraaifontein
  - King Edward VIII; Department of Haematology, KwaKhangela
- Spain (11):
  - Hospital Universitario Puerta del Mar; Servicio de Hematologia, Cadiz, Cadiz
  - Hospital del Mar; Servicio de Hematologia, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Duran i Reynals; Servicio de Hematologia, Barcelona
  - Hospital Universitario de la Princesa; Servicio de Hematologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen de Arrixaca; Servicio de Hematologia, Murcia
  - Hospital Clinico Universitario de Salamanca;Servicio de Hematologia, Salamanca
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
- Thailand (3):
  - National Cancer Inst., Bangkok
  - Siriraj Hospital; Division of Hematology, Department of Medicine, Bangkok
  - Srinagarind Hospital, Khon Kaen Uni ; Dept of Medicine, Khon Kaen
- Turkey (Türkiye) (5):
  - Adana Baskent University Hospital; Medical Oncology, Adana
  - Istanbul University Cerrahpasa Medical Faculty; Hematology Department, Istanbul
  - Bilim University School of Medicine; Hematology, Istanbul
  - Dokuz Eylul Uni ; Hematology, Izmir
  - Ege Uni Medical School; Hematology, Izmir
- United Kingdom (7):
  - Ninewells Hospital & Medical School; Ward 34, Dundee
  - Maidstone & Tonbridge Wells Hospital; Kent Oncology Center, Maidstone
  - Derriford Hospital; Department of Haematology, Plymouth
  - Queen's Hospital; Oncology, Romford
  - Southampton General Hospital, Southampton
  - Pinderfields General Hospital; Dept of Haematology, Wakefield
  - New Cross Hospital; Dept. Of Haematology, Wolverhampton

REFERENCES:
- [Derived] Davies A, Merli F, Mihaljevic B, Mercadal S, Siritanaratkul N, Solal-Celigny P, Boehnke A, Berge C, Genevray M, Zharkov A, Dixon M, Brewster M, Barrett M, MacDonald D. Efficacy and safety of subcutaneous rituximab versus intravenous rituximab for first-line treatment of follicular lymphoma (SABRINA): a randomised, open-label, phase 3 trial. Lancet Haematol. 2017 Jun;4(6):e272-e282. doi: 10.1016/S2352-3026(17)30078-9. Epub 2017 May 2. PMID 28476440
- [Derived] Davies A, Merli F, Mihaljevic B, Siritanaratkul N, Solal-Celigny P, Barrett M, Berge C, Bittner B, Boehnke A, McIntyre C, Macdonald D. Pharmacokinetics and safety of subcutaneous rituximab in follicular lymphoma (SABRINA): stage 1 analysis of a randomised phase 3 study. Lancet Oncol. 2014 Mar;15(3):343-52. doi: 10.1016/S1470-2045(14)70005-1. Epub 2014 Feb 10. PMID 24521993
- [Derived] Mao CP, Brovarney MR, Dabbagh K, Birnbock HF, Richter WF, Del Nagro CJ. Subcutaneous versus intravenous administration of rituximab: pharmacokinetics, CD20 target coverage and B-cell depletion in cynomolgus monkeys. PLoS One. 2013 Nov 12;8(11):e80533. doi: 10.1371/journal.pone.0080533. eCollection 2013. PMID 24265828
- [Derived] Shpilberg O, Jackisch C. Subcutaneous administration of rituximab (MabThera) and trastuzumab (Herceptin) using hyaluronidase. Br J Cancer. 2013 Sep 17;109(6):1556-61. doi: 10.1038/bjc.2013.371. Epub 2013 Sep 3. PMID 24002601

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening/baseline tests were performed within 28 days before randomization. Randomization was centralized in a 1:1 fashion using the Pocock and Simon dynamic randomization algorithm. The study was conducted in 2 stages: Stage I & II. All participants irrespective of the treatment period completion commenced follow-up period in both Stage I and II.
Groups:
- Stage I: Rituximab IV + Chemotherapy (CHOP/CVP): Eight cycles of rituximab intravenous (IV) infusion (375 milligrams per square meter [mg/m^2]; rituximab induction) in combination with up to 8 cycles of cyclophosphamide, doxorubicin, vincristine, prednisolone (CHOP) or cyclophosphamide, vincristine, prednisolone (CVP) chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least partial response (PR) during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
- Stage I: Rituximab SC + Chemotherapy (CHOP/CVP): First cycle of rituximab IV (375 mg/m^2) + 7 cycles of rituximab subcutaneously (SC) (1400 milligrams [mg]; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
- Stage II: Rituximab IV + Chemotherapy (CHOP/CVP): Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
- Stage II: Rituximab SC + Chemotherapy (CHOP/CVP): First cycle of rituximab IV (375 mg/m^2) + 7 cycles of rituximab SC (1400 mg; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
Period: Stage I
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP) | Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage II: Rituximab SC + Chemotherapy (CHOP/CVP)
Started | 64 | 63 | 0 (Different participants were randomized into different stages of the study.) | 0 (Different participants were randomized into different stages of the study.)
Completed | 46 (Participants completed treatment period.) | 46 (Participants completed treatment period.) | 0 | 0
Not Completed | 18 | 17 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0
Not completed — Adverse Event | 5 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Disease Progression | 9 | 7 | 0 | 0
Period: Stage 2
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP) | Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage II: Rituximab SC + Chemotherapy (CHOP/CVP)
Started | 0 (Different participants were randomized into different stages of the study.) | 0 (Different participants were randomized into different stages of the study.) | 141 | 142
Completed | 0 | 0 | 100 (Participants completed treatment period.) | 92 (Participants completed treatment period.)
Not Completed | 0 | 0 | 41 | 50
Not completed — Disease Progression | 0 | 0 | 16 | 21
Not completed — Lack of Efficacy | 0 | 0 | 4 | 2
Not completed — Physician Decision | 0 | 0 | 5 | 7
Not completed — Adverse Event | 0 | 0 | 5 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 4
Not completed — Death | 0 | 0 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all participants who were randomized into study irrespective whether they received study drug or not.
Groups:
- Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP): Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
- Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP): First cycle rituximab IV infusion (375 mg/m^2) + 7 cycles of rituximab SC 1400 mg in combination with up to 8 cycles of CHOP or CVP chemotherapy administered every 3 weeks. Participants achieving at least PR entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
- Total: Total of all reporting groups
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP) | Total
Number analyzed (Participants) | 205 | 205 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (12.69) [28 to 86] | 56.1 (12.66) [28 to 85] | 56.5 (12.67) [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 120 | 219
  Male | 106 | 85 | 191

OUTCOME MEASURES:

1. Primary Outcome: Stage I: Trough Serum Concentrations (Ctrough) of IV and SC Rituximab
Time Frame: Stage I: Cycle (Cy) 7 Day (D) 21 (within 2 hours predose on Cy8) of induction treatment (1 Cy=3 weeks)
Population: Stage I pharmacokinetic (PK) evaluable population comprised all participants with data for Ctrough available at Cycle 7 and/or observed area under the serum concentration-time curve (AUC) available at Cycle 7. Participants were analyzed as per treatment received. Number of participants analyzed = participants analyzed for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Stage I: Rituximab IV + Chemotherapy (CHOP/CVP): Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
- Stage I: Rituximab SC + Chemotherapy (CHOP/CVP): First cycle of rituximab IV (375 mg/m^2) + 7 cycles of rituximab subcutaneously (SC) (1400 mg; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 48 | 54
micrograms per milliliter (mcg/mL) | 83.1 (36.7) | 134.6 (43.2)
Statistical Analysis 1: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Non-Inferiority or Equivalence — Non-inferior Ctrough in SC formulation was demonstrated, if the lower bound of 90% confidence interval (CI) was above 0.8; Geometric mean ratio = 1.62, 90% CI 2-sided [1.36 to 1.94] — Geometric mean ratio adjusted for tumor load at baseline

2. Primary Outcome: Stage II: Percentage of Participants With Overall Response at the End of Induction Treatment Assessed Using International Working Group Response Criteria for Non-Hodgkin Lymphoma (NHL)
Description: Overall Response comprised complete response (CR), CR unconfirmed (CRu), or PR. A participant was defined as a responder if they sustained a CR, CRu or PR at the end of induction treatment. Response assessment was based on clinical examination and computed tomography (CT) scans. Assessment of tumor response was performed according to the International Working Group response criteria for NHL. CR: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CRu: CR along with regression in lymph node mass by more than (>) 75% in the sum of the products of greatest diameters (SPD); PR: Greater than or equal to (≥) 50% decrease in SPD of 6 largest dominant nodes or nodal masses. The 95% CI was estimated for one sample binomial using Pearson-Clopper.
Time Frame: Stage II: Baseline up to end of induction treatment Cy8 (24 weeks) (1 Cy=3 weeks)
Population: Stage II ITT Population included all participants who were randomized in Stage II irrespective whether they received study drug or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Stage II: Rituximab IV + Chemotherapy (CHOP/CVP): Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
- Stage II: Rituximab SC + Chemotherapy (CHOP/CVP): First cycle of rituximab IV infusion (375 mg/m^2) + 7 cycles of rituximab SC (1400 mg; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months.
Arm/Group | Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 141 | 142
percentage of participants | 85.1 [78.1 to 90.5] | 80.3 [72.8 to 86.5]
Statistical Analysis 1: Comparison: Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.2835, Chi-squared; Difference in response rates = -4.82, 95% CI 2-sided [-14.0 to 4.4] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.38 to 1.33]

3. Secondary Outcome: Stage I: Percentage of Participants With Overall Response at the End of Induction Treatment Assessed Using International Working Group Response Criteria for NHL
Description: Overall Response comprised CR, CRu, or PR. A participant was defined as a responder if they sustained a CR, CRu or PR at the end of induction treatment. Response assessment was based on clinical examination and CT scans. Assessment of tumor response was performed according to the International Working Group response criteria for NHL. CR: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CRu: CR along with regression in lymph node mass by >75% in the SPD; PR: ≥50% decrease in SPD of 6 largest dominant nodes or nodal masses. The 95% CI was estimated for one sample binomial using Pearson-Clopper.
Time Frame: Stage I: Baseline up to end of induction treatment Cy8 (24 weeks) (1 Cy=3 weeks)
Population: Stage I ITT Population included all participants who were randomized in Stage I irrespective whether they received study drug or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 64 | 63
percentage of participants | 82.8 [71.3 to 91.1] | 90.5 [80.4 to 96.4]
Statistical Analysis 1: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.2047, Chi-squared; Difference in response rates = 7.66, 95% CI 2-sided [-5.0 to 20.3] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.68 to 5.71]

4. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants With Overall Response at the End of Induction Treatment Assessed Using International Working Group Response Criteria for NHL
Description: Overall Response comprised of CR, CRu, or PR. A participant was defined as a responder if they sustained a CR, CRu or PR at the end of induction treatment. Response assessment was based on clinical examination and CT scans. Assessment of tumour response was performed according to the International Working Group response criteria for NHL. CR: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CRu: CR along with regression in lymph node mass by >75% in SPD; PR: ≥50% decrease in SPD of 6 largest dominant nodes or nodal masses. The 95% CI for the response rates was estimated for one sample binomial using Pearson-Clopper.
Time Frame: Stage I and II: Baseline up to end of induction treatment Cy8 (24 weeks) (1 Cy=3 weeks)
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
percentage of participants | 84.9 [79.2 to 89.5] | 84.4 [78.7 to 89.1]
Statistical Analysis 1: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.8911, Chi-squared; Difference in response rates = -0.49, 95% CI 2-sided [-7.7 to 6.8] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson
Statistical Analysis 2: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.56 to 1.65]

5. Secondary Outcome: Stage I: Percentage of Participants With Complete Response at the End of Induction Treatment Assessed Using International Working Group Response Criteria for NHL
Description: Complete Response was comprised CR and CRu. A participant was defined as a responder if they sustained a CR or CRu at the end of induction treatment. Response assessment was based on clinical examination and CT scans. Assessment of tumor response was performed according to the International Working Group response criteria for NHL. CR: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CRu: CR along with regression in lymph node mass by >75% in SPD. The 95% CI for the response rates was estimated for one sample binomial using Pearson-Clopper.
Time Frame: Stage I: Baseline up to end of induction treatment Cy8 (24 weeks) (1 Cy=3 weeks)
Population: Stage I ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 64 | 63
percentage of participants | 25.0 [15.0 to 37.4] | 42.9 [30.5 to 56.0]
Statistical Analysis 1: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.0335, Chi-squared; Difference in CRR = 17.86, 95% CI 2-sided [0.8 to 35.0] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.06 to 4.78]

6. Secondary Outcome: Stage II: Percentage of Participants With Complete Response at the End of Induction Treatment Assessed Using International Working Group Response Criteria for NHL
Description: Complete Response comprised of CR and CRu. A participant was defined as a responder if they sustained a CR or CRu at the end of induction treatment. Response assessment was based on clinical examination and CT scans. Assessment of tumor response was performed according to the International Working Group response criteria for NHL. CR: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CRu: CR along with regression in lymph node mass by >75% in SPD. The 95% CI for the response rates was estimated for one sample binomial using Pearson-Clopper.
Time Frame: Stage II: Baseline up to end of induction treatment Cy8 (24 weeks) (1 Cy=3 weeks)
Population: Stage II ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 141 | 142
percentage of participants | 34.8 [26.9 to 43.2] | 28.2 [20.9 to 36.3]
Statistical Analysis 1: Comparison: Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.2331, Chi-squared; Difference in response rates = -6.58, 95% CI 2-sided [-17.8 to 4.6] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.44 to 1.22]

7. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants With Complete Response at the End of Induction Treatment Assessed Using International Working Group Response Criteria for NHL
Description: as for outcome 6
Time Frame: Stage I and II: Baseline up to end of induction treatment Cy8 (24 weeks) (1 Cy=3 weeks)
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
percentage of participants | 31.7 [25.4 to 38.6] | 32.2 [25.9 to 39.1]
Statistical Analysis 1: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.9157, Chi-squared; Difference in response rates = 0.49, 95% CI 2-sided [-8.8 to 9.8] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.66 to 1.51]

8. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants With Complete Response at the End of Maintenance Treatment Assessed Using International Working Group Response Criteria for NHL
Description: as for outcome 6
Time Frame: Stage I and II: Baseline up to 57 days after last maintenance dose (last maintenance dose: maintenance Cy12/Study Cy20 [30 months]) (up to data cutoff of 31 Oct 2017 [up to 6 years]) (1 Cy=8 weeks)
Population: ITT population; only participants who entered the maintenance phase and received at least 1 cycle of rituximab maintenance treatment from Cycle 9 to Cycle 20 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 178 | 172
percentage of participants | 57.9 [50.3 to 65.2] | 50.6 [42.9 to 58.3]
Statistical Analysis 1: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.1715, Chi-squared; Difference in response rates = -7.28, 95% CI 2-sided [-18.0 to 3.5] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.52 to 1.22]

9. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants With Overall Response at the End of Maintenance Treatment Assessed Using International Working Group Response Criteria for NHL
Description: Overall Response comprised of CR, CRu, or PR . A participant was defined as a responder if they sustained a CR, CRu or PR at the end of induction treatment. Response assessment was based on clinical examination and CT scans. Assessment of tumor response was performed according to the International Working Group response criteria for NHL. CR: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CRu: CR along with regression in lymph node mass by >75% in SPD. The 95% CI for the response rates was estimated for one sample binomial using Pearson-Clopper.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 178 | 172
percentage of participants | 78.1 [71.3 to 83.9] | 77.9 [71.0 to 83.9]
Statistical Analysis 1: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.9671, Chi-squared; Difference in response rates = -0.18, 95% CI 2-sided [-9.2 to 8.8] — The 95% CI for the difference in response rates was estimated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.60 to 1.64]

10. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants With Disease Progression/Relapse or Death
Description: Disease progression: ≥50% increase from nadir in the SPD of any previously identified abnormal node or appearance of any new lesion during or at the end of therapy or ≥50% increase in the greatest diameter of any previously identified node >1 cm in its short axis or in the SPD of more than one node. Baseline, D1 of all cycles (Cy 1-20) (1 Cy=3 weeks for Cy1-8 & 8 weeks for Cy9-20), at early withdrawal, at follow-up, every 12 weeks for 96 weeks or until documented disease progression/relapse or death (up to median of 27 months; up to data cutoff of 31 Oct 2017 [up to 6 years])
Time Frame: Baseline up to disease progression or death up to data cutoff of 31 Oct 2017 (up to 6 years) (See detailed timeframe in Outcome Measure description)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
percentage of participants | 34.6 | 31.7

11. Secondary Outcome: Stage I and II (Pooled): Progression-Free Survival (PFS) Assessed Using International Working Group Response Criteria for NHL
Description: PFS was defined as the time from randomization to disease progression/relapse or death due to any cause. If the specified event (disease progression/relapse, death) did not occur, PFS was censored at the last tumor assessment date showing no disease progression, either during treatment or follow-up. Disease progression: ≥50% increase from nadir in the SPD of any previously identified abnormal node or appearance of any new lesion during or at the end of therapy or ≥50% increase in the greatest diameter of any previously identified node >1 cm in its short axis or in the SPD of more than one node. PFS analysis was performed using Kaplan - Meier curves. Baseline, D1 of all cycles (Cy 1-20) (1 Cy=3 weeks for Cy1-8 & 8 weeks for Cy9-20), at early withdrawal, at follow-up, every 12 weeks for 96 weeks or until documented disease progression/relapse or death (up to median of 27 months; up to data cutoff of 31 Oct 2017 [up to 6 years])
Time Frame: as for outcome 10
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
days | NA [NA to NA] — Data for upper limit of 95% CI were not reached due to low number (<50%) of participants with event of interest. | NA [NA to NA] — Data for median and corresponding 95% CI were not reached due to low number (<50%) of participants with event of interest.
Statistical Analysis 1: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.5526, Wald test; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.64 to 1.26]

12. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants With Disease Progression/Relapse, New Anti-Lymphoma Treatment or Death Assessed Using International Working Group Response Criteria for NHL
Description: Disease progression: ≥50% increase from nadir in the SPD of any previously identified abnormal node or appearance of any new lesion during or at the end of therapy or ≥50% increase in the greatest diameter of any previously identified node >1 cm in its short axis or in the SPD of more than one node. Baseline, D1 of all cycles (Cy 1-20) (1 Cy=3 weeks for Cy1-8 & 8 weeks for Cy9-20), at early withdrawal, at follow-up, every 12 weeks for 96 weeks or until documented disease progression/relapse or death (up to a median of 27 months; up to data cutoff of 31 Oct 2017 [up to 6 years])
Time Frame: as for outcome 10
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
percentage of participants | 36.1 | 35.1

13. Secondary Outcome: Stage I and II (Pooled): Event-Free Survival Assessed Using International Working Group Response Criteria for NHL
Description: Event-free survival was defined as the time from randomization to disease progression/relapse, death or initiation of new NHL therapy. If the specified event (progression/relapse, death or new anti-lymphoma treatment) did not occur, event-free survival was censored at the last tumor assessment date either during treatment or follow up. Event-free survival analysis was performed using Kaplan-Meier curves. Baseline, D1 of all cycles (Cy 1-20) (1 Cy=3 weeks for Cy1-8 & 8 weeks for Cy9-20), at early withdrawal, at follow-up, every 12 weeks for 96 weeks or until documented disease progression/relapse or death (up to a median of 27 months; up to data cutoff of 31 Oct 2017 [up to 6 years])
Time Frame: as for outcome 10
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
days | NA [2126 to NA] — Data for upper limit of 95% CI was not reached due to low number (<50%) of participants with event of interest. | NA [NA to NA] — Data for median and upper limit of 95% CI were not reached due to low number (<50%) of participants with event of interest.
Statistical Analysis 1: Comparison: Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; p = 0.9115, Wald test; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.71 to 1.36]

14. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline up to death (up to data cutoff of 31 Oct 2017 [up to 6 years])
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
percentage of participants | 12.7 | 8.8

15. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without event were censored at the time of last follow-up information for survival, ie, at the last time known to be alive.
Time Frame: Baseline up to death (up to data cutoff of 31 Oct 2017 [up to 6 years])
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 205 | 205
days | NA [NA to NA] — Data for median and corresponding 95% CI were not reached due to low number (<10%) of participants with event of interest. | NA [NA to NA] — Data for median and corresponding 95% CI were not reached due to low number (<10%) of participants with event of interest.

16. Secondary Outcome: Stage I: Observed Area Under the Serum Concentration-Time Curve (AUC) of Rituximab
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Predose (within 2 hr) and 24 hrs postdose on Cy 7 (D1,3,7,15), predose (0 hr) on Cy 8 D1 (1 Cy=3 weeks); additionally within 15 minutes after end of infusion (infusion duration=30 minutes) on Cy 7 D1 for rituximab IV (up to data cutoff of 11 Apr 2012 [up to 26 months])
Time Frame: Stage I (Induction): Predose (within 2 hour [hr]) up to data cutoff of 11 Apr 2012 [up to 26 months]) (See detailed timeframe in Outcome Measure description)
Population: Stage I PK evaluable population. Here, number of participants analyzed = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 58 | 55
mcg*day/mL | 2734.21 (32.51) | 3778.93 (37.59)
Statistical Analysis 1: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); The ratio of observed rituximab serum was determined as AUC SC/AUC IV during Cycle 7 of induction treatment; Test type: Superiority or Other; Geometric mean ratio = 1.38, 90% CI 2-sided [1.24 to 1.53]

17. Secondary Outcome: Stage I: Maximum Serum Concentrations (Cmax) of IV and SC Rituximab
Description: Predose (within 2 hr) and 24 hrs postdose on Cy7 (D1,3,7,15), predose (0 hr) on Cy8 D1 (1 Cy=3 weeks); additionally within 15 minutes after end of infusion (infusion duration=30 minutes) on Cy7 D1 for rituximab IV (up to data cutoff of 11 Apr 2012 [up to 26 months])
Time Frame: Stage I (Induction): Predose (within 2hr) up to data cutoff of 11 Apr 2012 [up to 26 months]) (See detailed timeframe in Outcome Measure description)
Population: Stage 1 PK Evaluable Population. Here, number of participants analyzed = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 58 | 59
mcg/mL | 250.63 (19.66) | 236.82 (31.45)
Statistical Analysis 1: Comparison: Stage I: Rituximab IV + Chemotherapy (CHOP/CVP) vs Stage I: Rituximab SC + Chemotherapy (CHOP/CVP); Test type: Superiority or Other; Geometric mean ratio = 0.941, 95% CI 2-sided [0.872 to 1.015]

18. Secondary Outcome: Stage I and II (Pooled): Ctrough of Rituximab at Each Induction Treatment Cycle
Description: Stage I and II (Induction): Rituximab IV: Predose (within 2 hr) on D1 of Cy1-8 (1 Cy=3 weeks & 4 weeks for Cy8); Rituximab SC: Predose (within 2 hr) on D1 of Cy1 & Cy3-8 (1 Cy=3 weeks and 4 weeks for Cy8), predose (within 2 hr) on D0 of Cy2 (up to data cutoff of 31 Oct 2013 [up to 32 months])
Time Frame: Stage I and II (Pooled): Predose (within 2hr) up to data cutoff of 31 Oct 2013 [up to 32 months]) (See detailed timeframe in Outcome Measure description)
Population: ITT Population. Here, number of participants analyzed = participants evaluable for the outcome measure. Here "n" = number of participants evaluable for this outcome measure at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 198 | 193
mcg/mL
  Cycle 1 (n = 198, 193) | 14.00 (157.53) | 12.88 (189.70)
  Cycle 2 (n = 197, 190) | 30.13 (145.36) | 40.00 (124.50)
  Cycle 3 (n = 192, 190) | 45.25 (110.35) | 63.83 (101.83)
  Cycle 4 (n = 186, 185) | 54.06 (108.90) | 81.71 (92.28)
  Cycle 5 (n = 185, 185) | 64.68 (89.90) | 98.00 (71.91)
  Cycle 6 (n = 187, 180) | 71.02 (87.60) | 109.56 (58.74)
  Cycle 7 (n = 183, 172) | 78.31 (77.76) | 120.75 (55.60)
  Cycle 8 (n = 52, 54) | 77.60 (70.53) | 131.48 (50.20)

19. Secondary Outcome: Stage I and II (Pooled): Ctrough of Rituximab at Each Maintenance Treatment Cycle
Description: Stage I and II (maintenance): D29 of Cy8 (induction; 1 Cy=4 weeks), predose (within 2 hr) on D1 of Cy9 to 19 (maintenance Cy1 to 12 [1 Cy=8 weeks]; up to data cutoff of 11 Jan 2016 [up to 6 years])
Time Frame: Stage I and II (maintenance): Predose (within 2hr) up to data cutoff of 11 Jan 2016 [up to 6 years]) (See detailed timeframe in Outcome Measure description)
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 174 | 170
mcg/mL
  Cycle 8 (n = 174, 170) | 37.69 (94.30) | 61.31 (65.52)
  Cycle 9 (n = 171, 168) | 30.35 (75.03) | 49.47 (81.23)
  Cycle 10 (n = 164, 160) | 28.44 (84.64) | 47.27 (73.03)
  Cycle 11 (n = 164, 157) | 28.77 (65.28) | 46.70 (66.80)
  Cycle 12 (n = 160, 150) | 28.80 (56.97) | 44.72 (68.74)
  Cycle 13 (n = 157, 150) | 28.84 (54.04) | 44.32 (67.67)
  Cycle 14 (n = 153, 147) | 28.09 (55.61) | 43.32 (67.97)
  Cycle 15 (n = 148, 143) | 28.19 (52.69) | 44.11 (67.92)
  Cycle 16 (n = 150, 145) | 28.05 (57.19) | 42.96 (64.32)
  Cycle 17 (n = 149, 143) | 28.24 (57.51) | 42.82 (65.67)
  Cycle 18 (n = 143, 132) | 28.59 (62.06) | 44.79 (68.56)
  Cycle 19 (n = 138, 131) | 27.75 (78.26) | 43.69 (69.02)

20. Secondary Outcome: Stage I and II (Pooled): Rituximab Levels 12 Weeks, 24 Weeks, and 36 Weeks After the Last Rituximab Administration
Time Frame: 12 weeks, 24 weeks, and 36 weeks after the last rituximab administration (up to data cutoff of 11 Jan 2016 [up to 6 years])
Population: Safety Analysis Population included all participants who received at least one dose of rituximab, either IV or SC. Participants were analyzed as treated. Here, number of participants analyzed = participants evaluable for the outcome measure. Here "n" = number of participants evaluable for this outcome measure at specified timepoint.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 117 | 118
mcg/mL
  Week 12: Follow-up Visit 1 (n = 117, 118) | 15.60 [0.70 to 80.40] | 22.35 [0.65 to 107.00]
  Week 24: Follow-up Visit 2 (n = 88, 96) | 2.89 [0.58 to 17.40] | 5.19 [0.69 to 62.10]
  Week 36: Follow-up Visit 3 (n = 38, 53) | 1.08 [0.52 to 51.40] | 2.02 [0.53 to 33.90]

21. Secondary Outcome: Percentage of Participants With B-Cell Depletion by Cycle for Induction Phase
Description: Depletion is defined as a cluster of differentiation (CD) 19 value <80 cells per cubic millimeter (cells/mm^3).
Time Frame: Stage I and II (induction): for rituximab IV - D1 of Cy 1 to 8 (1 Cy=3 weeks); for rituximab SC - D1 of Cy 1 and Cy 3 to 8, D0 of Cy 2
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 188 | 180
percentage of participants
  Cycle 1 Day 1 - Baseline (n=188, 168) | 51.6 | 54.8
  Cycle 2 Day 0 (n=183, 180) | 95.1 | 95.0
  Cycle 3 Day 1 (n=175, 175) | 99.4 | 99.4
  Cycle 4 Day 1 (n=178, 180) | 99.4 | 100.0
  Cycle 5 Day 1 (n=179, 176) | 100.0 | 100.0
  Cycle 6 Day 1 (n=173, 175) | 100.0 | 100.0
  Cycle 7 Day 1 (n=178, 173) | 100.0 | 100.0
  Cycle 8 Day 1 (n=175, 174) | 100.0 | 100.0

22. Secondary Outcome: Percentage of Participants With B-Cell Depletion by Cycle for Maintenance Phase
Description: Depletion is defined as a CD19 value <80 cells/mm^3.
Time Frame: Stage I and II (maintenance): D1 of Cy 9 to 20 (1 Cy=8 weeks) (up to data cutoff of 11 Jan 2016 [up to 6 years])
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 170 | 164
percentage of participants
  Cycle 9 Day 1 (n=170, 161) | 99.4 | 100.0
  Cycle 10 Day 1 (n=165, 164) | 99.4 | 100.0
  Cycle 11 Day 1 (n=158, 158) | 99.4 | 100.0
  Cycle 12 Day 1 (n=151, 146) | 100.0 | 100.0
  Cycle 13 Day 1 (n=149, 143) | 100.0 | 100.0
  Cycle 14 Day 1 (n=152, 143) | 100.0 | 100.0
  Cycle 15 Day 1 (n=149, 140) | 100.0 | 100.0
  Cycle 16 Day 1 (n=142, 141) | 100.0 | 100.0
  Cycle 17 Day 1 (n=145, 142) | 100.0 | 100.0
  Cycle 18 Day 1 (n=141, 140) | 100.0 | 100.0
  Cycle 19 Day 1 (n=140, 138) | 100.0 | 100.0
  Cycle 20 Day 1 (n=139, 134) | 100.0 | 100.0

23. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants Positive for Human Anti-Chimeric Antibodies (HACAs) to Rituximab
Description: Levels of HACA in serum were detected at Day 1 of each cycle up to Cycle 8 and at follow-up visit. Stage I and II: Baseline: pre-dose (72 hours prior) D1 of Cy1, Cy 3-20, D0 of Cy2 (1 Cy=3 weeks for Cy1-8 & 8 weeks for Cy9-20), post-baseline: every 12 weeks after last rituximab administration until 96 weeks (a median of 27 months; up to data cutoff of 11 Jan 2016 [up to 6 years])
Time Frame: Stage I and II: Baseline, post-baseline (See detailed timeframe in Outcome Measure description)
Population: Safety Analysis Population: included 6 participants who were randomized under Rituximab SC arm but withdrew after Cy1 and then analyzed under Rituximab IV arm. Here, number of participants analyzed = participants evaluable for the outcome measure. Here "n" = number of participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 208 | 197
percentage of participants
  Baseline (n=208, 191) | 5.8 | 2.6
  Post-Baseline (n=206, 197) | 1.5 | 2.0

24. Secondary Outcome: Stage I and II (Pooled): Percentage of Participants Positive for Human Anti-Human Antibodies (HAHAs) to Rituximab
Description: Levels of HAHA in serum were detected at Day 1 of each cycle up to Cycle 8 and at follow-up visit. Stage I and II: Baseline: pre-dose (72 hours prior) D1 of Cy1, Cy 3-20, D0 of Cy2 (1 Cy=3 weeks for Cy1-8 & 8 weeks for Cy9-20), post-baseline: every 12 weeks after last rituximab administration until 96 weeks (a median of 27 months; up to data cutoff of 11 Jan 2016 [up to 6 years])
Time Frame: Stage I and II: Baseline, post-baseline (See detailed timeframe in Outcome Measure description)
Population: Safety Analysis Population. Here, number of participants analyzed = participants evaluable for the outcome measure. Here "n" = number of participants evaluable for this outcome measure at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Number analyzed (Participants) | 68 | 197
percentage of participants
  Baseline (n=68, 188) | 10.3 | 11.2
  Post-Baseline (n=66, 197) | 7.6 | 13.2

25. Secondary Outcome: Stage I and II (Pooled): Percentage of Responses Showing Time Saved of Staff as Per Physician/Nurse Opinions With Each Administration of Rituximab SC as Compared to Rituximab IV at the End of Cy 8, 15 and 20
Description: All investigator physicians and nurses involved in this study were asked to provide the staff time that could be saved with each administration of rituximab SC as compared with rituximab IV to participants in routine practice afetr Cy 8, 15, 20 and categorized as less than (<) 1 hr, at least 1 hr but <2 hrs, at least 2 hrs but <3 hrs, at least 3 hrs but <4 hrs, >/=4 hrs. Staff were asked not to consider the time needed for the first IV administration. Analysis was done in all participants to show a comparison on the time saved by staffs when administered via SC and IV.
Time Frame: After Cycle 8 of induction treatment (24 weeks) and during the maintenance part of the study after 12 months (i.e., Cycle 15), and after the end of the maintenance treatment, (i.e., Cycle 20) (1 Cycle=4 weeks for Cycle 8 and 8 weeks for Cycles 15 and 20)
Population: as for outcome 18
Measure: Number; unit: percentage of responses
Groups:
- All Participants: Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP): First cycle rituximab IV infusion (375 mg/m^2) + 7 cycles of rituximab SC 1400 mg in combination with up to 8 cycles of CHOP or CVP chemotherapy administered every 3 weeks. Participants achieving at least PR entered rituximab SC (1400 mg) maintenance therapy once every 8 weeks for 24 months. Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP): Eight cycles of rituximab IV infusion (375 mg/m^2; rituximab induction) in combination with up to 8 cycles of CHOP or CVP chemotherapy (as per institutional practice) administered every 3 weeks. Participants achieving at least PR during induction, entered rituximab IV maintenance therapy (375 mg/m^2) once every 8 weeks for 24 months.
Arm/Group | All Participants
Number analyzed (Participants) | 166
percentage of responses
  After Cy8: <1 hour (n=166) | 11
  After Cy8: ≥1 to <2 hours (n=166) | 20
  After Cy8: ≥2 to <3 hours (n=166) | 35
  After Cy8: ≥3 to <4 hours (n=166) | 18
  After Cy8: ≥4 hours (n=166) | 16
  After Cy15: <1 hour (n=130) | 13
  After Cy15: ≥1 to <2 hours (n=130) | 17
  After Cy15: ≥2 to <3 hours (n=126) | 34
  After Cy15: ≥3 to <4 hours (n=130) | 14
  After Cy15: ≥4 hours (n=130) | 22
  After Cy20: <1 hour (n=126) | 14
  After Cy20: ≥1 to <2 hours (n=126) | 32
  After Cy20: ≥2 to <3 hours (n=126) | 21
  After Cy20: ≥3 to <4 hours (n=126) | 13
  After Cy20: ≥4 hours (n=126) | 19

26. Secondary Outcome: Percentage of Responses Who Showed Rituximab SC Formulation Convenient as Compared to Rituximab IV Formulation as Assessed by Physician/Nurse Opinion
Description: All investigator physicians and nurses involved in this study were asked to complete question i.e. "Which formulation of rituximab (SC or IV) do you think is more convenient?" based on their experience with the rituximab SC and IV formulations across all participants and presented as rituximab SC is much more convenient; rituximab SC is a little more convenient; both formulations are equally convenient; rituximab IV is a little more convenient; and rituximab IV is much more convenient.
Time Frame: as for outcome 25
Population: as for outcome 18
Measure: Number; unit: percentage of responses
Arm/Group | All Participants
Number analyzed (Participants) | 166
percentage of responses
  Cy8: Rituximab SC much more convenient (n=166) | 81
  Cy8: Rituximab SC little more convenient (n=166) | 13
  Cy8: Both formulations equally convenient (n=166) | 2
  Cy8: Rituximab IV little more convenient (n=166) | 4
  Cy8: Rituximab IV much more convenient (n=166) | 0
  Cy15: Rituximab SC much more convenient (n=130) | 88
  Cy15: Rituximab SC little more convenient (n=130) | 7
  Cy15: Both formulations equally convenient (n=130) | 5
  Cy15: Rituximab IV little more convenient (n=130) | 0
  Cy15: Rituximab IV much more convenient (n=130) | 0
  Cy20: Rituximab SC much more convenient (n=126) | 88
  Cy20: Rituximab SC little more convenient (n=126) | 9
  Cy20: Both formulations equally convenient (n=126) | 2
  Cy20: Rituximab IV little more convenient (n=126) | 1
  Cy20: Rituximab IV much more convenient (n=126) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to data cutoff date of 31 Oct 2017 (up to 6 years)
Description: Safety Analysis Population included all participants who received at least one dose of rituximab, either IV or SC. Safety Analysis Population included 6 participants who were randomized under Rituximab SC arm but withdrew after Cy1 and then analyzed under Rituximab IV arm.
Arm/Group | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP)
Serious Adverse Events (participants affected / at risk) | 76/210 | 74/197
Other Adverse Events (participants affected / at risk) | 187/210 | 186/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) (N=210) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP) (N=197)
Pneumonia (Infections and infestations) | 7 | 11
Neutropenic sepsis (Infections and infestations) | 4 | 1
Cystitis (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 3
Bacterial prostatitis (Infections and infestations) | 0 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Giardiasis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 12
Neutropenia (Blood and lymphatic system disorders) | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Oral lichen planus (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 6
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Coma hepatic (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Pelvic cyst (Reproductive system and breast disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 2
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Chronic hepatitis B (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Intestinal sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection fungal (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cognitive disorder (Nervous system disorders) | 2 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Bladder calculus removal (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage I and II: Rituximab IV + Chemotherapy (CHOP/CVP) (N=210) | Stage I and II: Rituximab SC + Chemotherapy (CHOP/CVP) (N=197)
Nausea (Gastrointestinal disorders) | 47 | 65
Constipation (Gastrointestinal disorders) | 55 | 50
Diarrhoea (Gastrointestinal disorders) | 35 | 34
Vomiting (Gastrointestinal disorders) | 27 | 29
Abdominal pain (Gastrointestinal disorders) | 25 | 29
Dyspepsia (Gastrointestinal disorders) | 14 | 16
Injection site erythema (General disorders) | 0 | 27
Fatigue (General disorders) | 38 | 42
Asthenia (General disorders) | 27 | 35
Pyrexia (General disorders) | 29 | 29
Chills (General disorders) | 18 | 16
Mucosal inflammation (General disorders) | 12 | 9
Chest pain (General disorders) | 7 | 14
Injection site pain (General disorders) | 0 | 16
Neutropenia (Blood and lymphatic system disorders) | 57 | 65
Anaemia (Blood and lymphatic system disorders) | 26 | 30
Leukopenia (Blood and lymphatic system disorders) | 23 | 13
Paraesthesia (Nervous system disorders) | 27 | 30
Neuropathy peripheral (Nervous system disorders) | 30 | 24
Dizziness (Nervous system disorders) | 15 | 16
Headache (Nervous system disorders) | 20 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 16 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 22
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 28
Erythema (Skin and subcutaneous tissue disorders) | 11 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 20
Rash (Skin and subcutaneous tissue disorders) | 14 | 20
Upper respiratory tract infection (Infections and infestations) | 26 | 30
Urinary tract infection (Infections and infestations) | 28 | 16
Nasopharyngitis (Infections and infestations) | 25 | 22
Bronchitis (Infections and infestations) | 15 | 15
Sinusitis (Infections and infestations) | 10 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 49
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 21
Insomnia (Psychiatric disorders) | 19 | 19
Abdominal pain upper (Gastrointestinal disorders) | 11 | 11
Stomatitis (Gastrointestinal disorders) | 11 | 12
Oedema peripheral (General disorders) | 13 | 10
Influenza like illness (General disorders) | 12 | 5
Conjunctivitis (Infections and infestations) | 12 | 9
Influenza (Infections and infestations) | 14 | 9
Pneumonia (Infections and infestations) | 4 | 12
Hypertension (Vascular disorders) | 13 | 12
Hypoaesthesia (Nervous system disorders) | 7 | 10
Anxiety (Psychiatric disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.